CLINICAL TRIAL: NCT03109262
Title: High Quality Imaging and Dosimetry of Yttrium-90 (90Y) SIRT Using a Digital PET/CT
Brief Title: Yttrium-90 (Y90) Glass Microspheres PET/CT in Imaging Patients With Liver Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrei Iagaru, Professor of Radiology (Nuclear Medicine), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-39332; NCI-2017-00463 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VAR0147 (Other: OnCore)
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Primary Malignant Liver Neoplasm
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — X-Rays; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Yttrium Y-90 PET/CT vs 99mTc-MAA SPECT/CT Scans (Experimental): All participants receive both Y-90 PET/CT vs 99mTc-MAA SPECT/CT Scans
  Interventions: Procedure: Computed Tomography (CT); Procedure: Positron Emission Tomography (PET); Device: 90-Yttrium (Y-90) Glass Microspheres; Diagnostic Test: Technetium 99mTc albumin aggregated (99mTc-MAA); Procedure: Single-photon emission computerized tomography (SPECT) scan

INTERVENTIONS:
Procedure: Computed Tomography (CT) — As part of PET/CT and SPECT/CT scans.
  Other Names: CAT; CAT Scan; Computed Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography; X-ray
Procedure: Positron Emission Tomography (PET) — As part of PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Device: 90-Yttrium (Y-90) Glass Microspheres — Radiolabel for PET/CT scan
  Other Names: TheraSphere
Diagnostic Test: Technetium 99mTc albumin aggregated (99mTc-MAA) — Radiolabel for 99mTc-MAA SPECT/CT Scan
  Other Names: 99mTc-MAA
Procedure: Single-photon emission computerized tomography (SPECT) scan — As part of SPECT/CT scan
  Other Names: SPECT Scan

SUMMARY:
This clinical trial studies how well yttrium-90 (Y90) glass microspheres positron emission tomography (PET)/computed tomography (CT) works in imaging patients with liver tumors . Images produced by PET/CT may provide better information about the distribution of particles, such as Y90 glass microspheres, delivered for selective internal radiation therapy (SIRT) as compared to regular medical care images useing technetium Tc-99m albumin-aggregated single photon emission computed tomography (SPECT)/CT images.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the image quality of yttrium-90 (Y90) microspheres PET/CT post SIRT images as compared to technetium Tc-99m albumin aggregated (99mTc MAA) SPECT/CT.

SECONDARY OBJECTIVES:

I. To determine the superior accuracy in both distribution and dosimetry of Y90 PET/CT post-SIRT imaging compared to 99mTc MAA planar and SPECT/CT imaging.

OUTLINE:

Immediately after standard of care SIRT, patients receive Y90 glass microspheres and undergo PET/CT over 30 minutes.

This study compares the experimental images to the regular medical care images in the same participant.

ELIGIBILITY:
Inclusion Criteria:

* Patient provides written informed consent
* Patient is referred for 90Y SIRT radioembolization of liver tumor(s)
* Patient is capable of complying with study procedures
* Patient is able to remain still for duration of imaging procedure (approximately 30 minutes total for digital PET/CT)

Exclusion Criteria:

* Patient is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duan H, Khalaf MH, Ferri V, Baratto L, Srinivas SM, Sze DY, Iagaru A. High quality imaging and dosimetry for yttrium-90 (90Y) liver radioembolization using a SiPM-based PET/CT scanner. Eur J Nucl Med Mol Imaging. 2021 Jul;48(8):2426-2436. doi: 10.1007/s00259-021-05188-4. Epub 2021 Jan 14. PMID 33443618

RESULTS

PARTICIPANT FLOW:
Groups:
- Yttrium Y-90 PET/CT vs 99mTc-MAA SPECT/CT Scans: All participants receive both Y-90 PET/CT vs 99mTc-MAA SPECT/CT Scans
  * Computed Tomography (CT): As part of PET/CT and SPECT/CT scans.
  * Positron Emission Tomography (PET): As part of PET/CT scan
  * Single-photon emission computerized tomography (SPECT) scan: As part of SPECT/CT scan
  * 90-Yttrium (Y-90) Glass Microspheres: Radiolabel for PET/CT scan
  * Technetium 99mTc albumin aggregated (99mTc-MAA): Radiolabel for 99mTc-MAA SPECT/CT Scan
Period: Overall Study
Arm/Group | Yttrium Y-90 PET/CT vs 99mTc-MAA SPECT/CT Scans
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Yttrium Y-90 PET/CT vs 99mTc-MAA SPECT/CT Scans
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Image Quality for 90-Y PET/CT Scans
Description: Image quality for 90Y PET/CT scan images was assessed relative to the expected image quality of Standard of Care (SoC) 99mTc-MAA SPECT/CT scans obtained from the same participant. Assessments were conducted at 5, 10, 15 and 20 minutes after infusion. Scans were assessed on a 1 to 5 Likert scale by 2 Nuclear Medicine physicians who were blinded to patient information. The Likert scale for image quality was established as follows:
  1. = Non-diagnostic
  2. = Suboptimal
  3. = Acceptable
  4. = Good
  5. = Excellent, equivalent to a SoC 99mTc-MAA SPECT/CT scan The scans for each individual participant at each timepoint was scored on the Likert scale, as determined by the 2 Nuclear Medicine physicians. The outcome is reported as the overall mean of the physician determinations for each time point, with standard deviation.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yttrium Y-90 PET/CT vs 99mTc-MAA SPECT/CT Scans
Number analyzed (Participants) | 42
units on a scale
  5 minutes | 3.56 (0.43)
  10 minutes | 4.63 (0.49)
  15 minutes | 4.89 (0.28)
  20 minutes | 4.93 (0.21)

2. Secondary Outcome: Radiopharmaceutical Dosimetry Accuracy for 90-Y PET/CT Scans and 99mTc-MAA SPECT/CT Scans
Description: Radiopharmaceutical dosimetry was assessed based on the numerical tumor-absorbed dose value in Gray as calculated by SurePlan (MIM Software Inc, Cleveland, Ohio). The outcome is reported as the median tumor-absorbed dose in Gray for each scan method (90Y PET/CT and 99mTc-MAA SPECT/CT), with standard deviation.
Time Frame: 1 day
Measure: Median (Standard Error); unit: Gray
Groups:
- Yttrium Y-90 PET/CT: All participants receive Y-90 PET/CT Scan
  Computed Tomography (CT): As part of PET/CT scan. Positron Emission Tomography (PET): As part of PET/CT scan
  90-Yttrium (Y-90) Glass Microspheres: Radiolabel for PET/CT scan
- 99mTc-MAA SPECT/CT Scans: All participants receive 99mTc-MAA SPECT/CT scan
  Computed Tomography (CT): As part of SPECT/CT scans. Single-photon emission computerized tomography (SPECT) scan: As part of SPECT/CT scan
  Technetium 99mTc albumin aggregated (99mTc-MAA): Radiolabel for 99mTc-MAA SPECT/CT Scan
Arm/Group | Yttrium Y-90 PET/CT | 99mTc-MAA SPECT/CT Scans
Number analyzed (Participants) | 42 | 42
Gray | 142.9 (99.7) | 118.9 (91.0)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Yttrium Y-90 PET/CT vs 99mTc-MAA SPECT/CT Scans
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT03109262/Prot_SAP_001.pdf
  • Informed Consent Form (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03109262/ICF_000.pdf